CLINICAL TRIAL: NCT00322374
Title: A Phase I Study of Ixabepilone in Combination With Epirubicin in Patients With Metastatic Breast Cancer
Brief Title: Phase I Combination w/ Epirubicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-104; Eudract No: 2005-004864-22
Record Dates: First submitted 2006-05-01; First posted 2006-05-05 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Epothilones; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 25 mg/m^2 Ixabepilone plus 75 mg/m^2 Epirubicin (Experimental): Participants received 25 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
  Interventions: Drug: Ixabepilone; Drug: Epirubicin
- 30 mg/m^2 Ixabepilone plus 75 mg/m^2 Epirubicin (Experimental): Participants received 30 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
  Interventions: Drug: Ixabepilone; Drug: Epirubicin
- 35 mg/m^2 Ixabepilone plus 75 mg/m^2 Epirubicin (Experimental): Participants received 35 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
  Interventions: Drug: Ixabepilone; Drug: Epirubicin

INTERVENTIONS:
Drug: Ixabepilone — Infusion, intravenous (IV), Cycle = 21 days. Dose escalation study.
  Other Names: IXEMPRA®; BMS-247550; Epothilone
Drug: Epirubicin — Infusion, intravenous (IV): 75 mg/m^2. Cycle = 21 days, up to 10 cycles or cumulative dose of 800 mg/m².

SUMMARY:
Tumor response information was obtained for all participants who received at least 2 cycles of study drug, underwent requisite baseline and on-treatment disease assessments and had at least one post-treatment assessment. Tumor response assessment in evaluable participants was done according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥18 years
* Histologically or cytologically confirmed diagnosis of metastatic breast cancer
* Measurable or nonmeasurable disease defined by Response Evaluation Criteria In Solid Tumors (RECIST)

Exclusion Criteria:

* Number of prior chemotherapy lines of treatment in the metastatic setting ≥2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Local Institution, Toulouse, France
- Local Institution, Milan, Italy

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2: Participants received 25 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
- Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2: Participants received 30 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
- Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2: Participants received 35 mg/m^2 Ixabepilone as a 3-hour IV infusion following a 3- to 5-minute IV infusion of 75 mg/m^2 epirubicin every 21 days.
Period: Enrollment
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 | All Participants
Started | 0 | 0 | 0 | 42
Completed | 0 | 0 | 0 | 42
Not Completed | 0 | 0 | 0 | 0
Period: Starting Dose
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 | All Participants
Started | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0
Not completed — Study Drug Toxicity | 4 | 0 | 0 | 0
Period: First Escalation
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 | All Participants
Started | 0 | 30 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 30 | 0 | 0
Not completed — Documented Disease Progression | 0 | 6 | 0 | 0
Not completed — Physician Decision | 0 | 12 | 0 | 0
Not completed — Study Drug Toxicity | 0 | 11 | 0 | 0
Not completed — Participant Request | 0 | 1 | 0 | 0
Period: Second Escalation
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 | All Participants
Started | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 6 | 0
Not completed — Physician Decision | 0 | 0 | 5 | 0
Not completed — Study Drug Toxicity | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 | Total
Number analyzed (Participants) | 6 | 30 | 6 | 42
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 6 | 24 | 5 | 35
  >=65 years | 0 | 6 | 1 | 7
Age, Continuous [Median (Full Range); unit: years] | 57.5 [48 to 61] | 57.5 [38 to 69] | 53.5 [33 to 68] | 57 [33 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 30 | 6 | 42
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 5 | 16 | 3 | 24
  Italy | 1 | 14 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose Limiting Toxicity (DLT)
Description: DLT: any of the following considered related to ixabepilone, epirubicin or combination occurring in Cycle 1: Absolute neutrophil count <500 cells/mm^3 for ≥7 consecutive days or febrile neutropenia of any duration;Grade(Gr)4 thrombocytopenia <25,000 cells/mm^3 or Gr3 w/bleeding requiring platelet transfusion;Any other drug-related Gr3/4 non-hematologic toxicity except Gr3 injection site reaction, fatigue, transient arthralgia/myalgia;Delayed recovery to Gr≤1 or baseline (except for alopecia) from toxicity related to treatment w/ ixabepilone + epirubicin delaying initiation of next cycle ≥3 wks
Time Frame: From Baseline to the end of Cycle 1 (Day 21)
Population: The evaluable participant population consisted of participants who met the minimum safety evaluation requirements of the study: participant received ≥1 dose of ixabepilone and epirubicin in Cycle 1, completed adequate safety evaluations, and was observed for ≥21 days following the first dose or the participant experienced DLT.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Participants with DLT:Grade 4 (severe) neutropenia | 1 | 1 | 2
  Total Participants with DLT | 1 | 1 | 2
  Participants without DLT | 5 | 5 | 4

2. Primary Outcome: Ixabepilone Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (R2PD)
Description: The MTD was the highest dose in which 0/6 or 1/6 participants experienced DLT with at least 2 out of no more than 6 participants experiencing DLT at the next higher dose level. The RP2D was based on the MTD and the assessment of any relevant chronic toxicity. To obtain further confidence in the RP2D, a total maximum of 30 evaluable participants were enrolled at the MTD.
Time Frame: Day 21 of Cycle 1
Population: The evaluable participant population consisted of participants who met the minimum safety evaluation requirements of the study: participant received ≥1 dose of ixabepilone and epirubicin in Cycle 1, completed adequate safety evaluations, and were observed for ≥21 days following the first dose or the participant experienced DLT.
Measure: Number; unit: mg^m2
Groups:
- All Participants With Measurable Disease and Tumor Response: All participants received Ixabepilone administered as a 3-hour IV infusion following a 3- to 5-minute IV infusion of Epirubicin every 21 days.
Arm/Group | All Participants With Measurable Disease and Tumor Response
Number analyzed (Participants) | 42
mg^m2
  MTD | 30
  R2PD | 30

3. Secondary Outcome: Number of Participants With Death, Adverse Events (AEs), Serious Adverse Events (SAEs), Grade 3/4 AEs, or AEs Leading to Discontinuation
Description: AEs and SAEs considered possibly, probably, or certainly related to study treatment, graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).SAE= any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization/prolongation of existing hospitalization, results in persistent/significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event
Time Frame: Evaluated continuously on study from Baseline to ≤30 days after the last dose of study drug.
Population: All participants who received at least 1 cycle of therapy were evaluable for safety; adverse events and other symptoms were graded according to CTCAE Version 3.0.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 30 | 6
participants
  Deaths (total) | 0 | 0 | 0
  Deaths within 30 days of last dose | 0 | 0 | 0
  AEs | 6 | 30 | 6
  SAEs | 2 | 8 | 1
  Grade 3/4 AEs | 6 | 28 | 6
  AEs leading to discontinuation of study treatment | 4 | 12 | 1

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Single-dose Ixabepilone
Description: Pharmacokinetics (PK) is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmax=maximum observed plasma concentration of single-dose ixabepilone administered with IV dose of epirubicin 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 120 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
ng/ml | 169.00 (44.42) | 217.86 (53.56) | 251.83 (48.56)

5. Secondary Outcome: Area Under the Curve, Extrapolated to Infinity (AUC[INF]) of Single-dose Ixabepilone
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. AUC(INF)=area under the plasma concentration-time curve from time zero extrapolated to infinite time of single-dose ixabepilone administered with IV dose of epirubicin 75 mg/m^2.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 120 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
ng·h/mL | 1760.42 (535.89) | 2072.43 (399.60) | 2100.56 (353.87)

6. Secondary Outcome: Terminal Half-life (T-Half) of Single-dose Ixabepilone
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. T-Half=terminal-phase elimination half-life in plasma of single-dose ixabepilone administered with IV dose of epirubicin 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 120 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
hours | 51.82 (15.47) | 34.07 (11.75) | 44.15 (18.41)

7. Secondary Outcome: Clearance (CLT) of Single-dose Ixabepilone
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. CLT= Total body clearance from plasma of single-dose ixabepilone administered with IV dose of epirubicin 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 120 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
L/h | 26.03 (5.45) | 24.62 (5.56) | 26.68 (2.83)

8. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Single-dose Ixabepilone
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Vss= Volume of distribution at steady-state of single-dose ixabepilone administered with IV dose of epirubicin 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 120 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
liters | 1331.65 (370.88) | 803.21 (292.09) | 1001.70 (317.23)

9. Secondary Outcome: Epirubicin Cmax
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmax=maximum observed plasma concentration of epirubicin administered IV 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 24 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 28 | 6
ng/ml | 3306.53 (2125.45) | 4139.00 (2598.19) | 4533.08 (2490.83)

10. Secondary Outcome: Epirubicin AUC(INF)
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. AUC(INF)=the area under the plasma concentration-time curve from time zero extrapolated to infinity of epirubicin administered IV 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 24 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 27 | 6
ng·h/mL | 2489.37 (1488.39) | 3132.67 (1685.32) | 2595.44 (1017.64)

11. Secondary Outcome: Epirubicin T-Half
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. T-Half=terminal-phase elimination half-life in plasma of epirubicin administered IV dose 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 24 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 27 | 6
hours | 13.61 (3.33) | 19.41 (6.31) | 15.55 (2.92)

12. Secondary Outcome: Epirubicin CLT
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. CLT= Total body clearance from plasma of epirubicin administered IV 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 24 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 27 | 6
L/h | 81.33 (70.84) | 53.85 (32.87) | 58.00 (38.82)

13. Secondary Outcome: Epirubicin Vss
Description: PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Vss= Volume of distribution at steady-state of epirubicin administered IV 75 mg/m^2, derived from plasma concentration versus time data.
Time Frame: From the start of the ixabepilone infusion on Day 1 to 24 hours after the first infusion.
Population: Participants who had received any treatment with ixabepilone and epirubicin and had adequate concentration profiles.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Number analyzed (Participants) | 6 | 27 | 6
liters | 912.83 (1500.018) | 750.24 (977.352) | 522.45 (657.97)

14. Secondary Outcome: Number Of Participants With A Best Overall Tumor Response of Complete Response, Partial Response, Stable Disease, And Progressive Disease
Description: Information on all tumor lesions was obtained at baseline by radiologic techniques, or if appropriate by physical examination (e.g. subcutaneous nodules). Measurable tumors were evaluated using Response Evaluation Criteria In Solid Tumors (RECIST) criteria, wherein complete response (CR) = disappearance of all target lesions; partial response (PR) = ≥30% decrease in the sum of the longest diameter of target lesions; progressive disease (PD)= ≥20% increase in the sum of the longest diameter of target lesions, and stable disease (SD) = small changes that do not meet above criteria.
Time Frame: From Baseline (up to 2 weeks prior to starting therapy) to the end Cycle 2
Population: Participants with measurable disease who received any treatment, as well as response evaluable participants. Evaluations were based on tumor measurements collected on the case report form using RECIST incorporating the use of target/non-target lesions.
Measure: Number; unit: participants
Groups:
- All Participants With Measurable Disease: Participants with measurable disease at baseline per RECIST
- All Response-evaluable Participants: Participants treated at the MTD with measurable disease at baseline per RECIST
Arm/Group | All Participants With Measurable Disease | All Response-evaluable Participants
Number analyzed (Participants) | 32 | 22
participants
  Complete Response | 0 | 0
  Partial Response | 18 | 9
  Stable Disease | 11 | 10
  Progressive Disease | 3 | 3

15. Secondary Outcome: Duration of Tumor Response
Description: Defined as the interval measured from the time that the measurement criteria are first met for CR or PR, whichever occurs first, until the date of documented progressive disease or death. CR= disappearance of all target lesions; PR= ≥30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Time (in months) when criteria for CR or PR are met (which ever occurs first) up to date of progressive disease.
Population: as for outcome 14
Measure: Median (Full Range); unit: months
Groups:
- All Participants With Measurable Disease and Tumor Response: All participants with measurable disease and with a best tumor response of either CR or PR.
- All Response-evaluable Participants: Participants treated at the MTD with a best response of either CR or PR.
Arm/Group | All Participants With Measurable Disease and Tumor Response | All Response-evaluable Participants
Number analyzed (Participants) | 18 | 9
months | 6.45 [1 to 17] | 6.4 [2 to 10]

16. Secondary Outcome: Number Of Participants With Tumor Response by Duration of Response Category
Description: Duration of response was defined as the interval measured from the time that the measurement criteria are first met for CR or PR, whichever occurs first, until the date of documented progressive disease or death; PR= ≥30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Time (in months) when criteria for CR or PR are met (which ever occurs first) up to date of progressive disease.
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | All Participants With Measurable Disease and Tumor Response | All Response-evaluable Participants
Number analyzed (Participants) | 18 | 9
participants
  Response Duration < 4 Months | 5 | 1
  Response Duration ≥4 Months | 13 | 8
  Response Duration ≥6 Months | 11 | 6

ADVERSE EVENTS:
Arm/Group | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2
Serious Adverse Events (participants affected / at risk) | 2/6 | 8/30 | 1/6
Other Adverse Events (participants affected / at risk) | 6/6 | 30/30 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 (N=6) | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 (N=30) | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 (N=6)
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 2 | 0
VOMITING (Gastrointestinal disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 0 | 2 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PYREXIA (General disorders) | 0 | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone 25 mg^m2 + Epirubicin 75 mg^m2 (N=6) | Ixabepilone 30 mg^m2 + Epirubicin 75 mg^m2 (N=30) | Ixabepilone 35 mg^m2 + Epirubicin 75 mg^m2 (N=6)
CONJUNCTIVITIS (Eye disorders) | 0 | 2 | 1
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 2 | 6 | 1
HAEMOGLOBIN DECREASED (Investigations) | 1 | 8 | 3
PLATELET COUNT DECREASED (Investigations) | 1 | 1 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 2 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 2 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 3 | 2
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 1
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 1 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0 | 0
HOT FLUSH (Vascular disorders) | 0 | 2 | 1
VENOUS INSUFFICIENCY (Vascular disorders) | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 3 | 0
HEADACHE (Nervous system disorders) | 2 | 6 | 1
AREFLEXIA (Nervous system disorders) | 1 | 3 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 9 | 2
DYSAESTHESIA (Nervous system disorders) | 0 | 5 | 1
HYPOREFLEXIA (Nervous system disorders) | 3 | 10 | 2
PARAESTHESIA (Nervous system disorders) | 5 | 15 | 3
SENSORY LOSS (Nervous system disorders) | 2 | 9 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 2 | 2
HYPERAESTHESIA (Nervous system disorders) | 0 | 3 | 0
CRANIAL NEUROPATHY (Nervous system disorders) | 0 | 0 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 | 2 | 1
NAUSEA (Gastrointestinal disorders) | 5 | 25 | 4
VOMITING (Gastrointestinal disorders) | 3 | 21 | 4
DIARRHOEA (Gastrointestinal disorders) | 0 | 7 | 3
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 5 | 2
STOMATITIS (Gastrointestinal disorders) | 0 | 5 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 10 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 2 | 1
GINGIVAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 3 | 0
ONYCHOMYCOSIS (Infections and infestations) | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 1 | 0 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 1 | 5 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 3 | 1
ANAEMIA (Blood and lymphatic system disorders) | 5 | 20 | 3
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 11 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 6 | 30 | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 21 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3 | 4 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
BARTHOLINITIS (Reproductive system and breast disorders) | 0 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 11 | 4
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 9 | 3
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 0 | 4 | 1
PYREXIA (General disorders) | 1 | 3 | 1
ASTHENIA (General disorders) | 4 | 16 | 2
HYPERTHERMIA (General disorders) | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.